CLINICAL TRIAL: NCT01604460
Title: Randomized Evaluation of the Use of Plastic Bags to Prevent Neonatal Hypothermia in Developing Countries-Part V
Brief Title: Evaluation of Use of Plastic Bags to Prevent Neonatal Hypothermia-Part V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Health System, Alabama (Other)
Responsible Party: Principal Investigator, Waldemar A. Carlo, MD, Edwin M. Dixon Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 010
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Hypothermia; Newborn
Keywords: Hypothermia; Newborn; Plastic bag; Resuscitation
MeSH Terms: conditions — Hypothermia | interventions — Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resuscitation-no plastic bag (Sham Comparator): Resuscitation per standard of care without a plastic bag
  Interventions: Procedure: Resuscitation-no plastic bag
- Resuscitation-torso bag (Active Comparator): Use of plastic bag covering the torso and lower extremities for temperature regulation during and after resuscitation for the first hour after birth
  Interventions: Procedure: Resuscitation with torso plastic bag

INTERVENTIONS:
Procedure: Resuscitation with torso plastic bag — Infant will be placed within 10 minutes of his birth into a plastic bag to his/her axillae and the bag will be folded and taped to itself to prevent it from covering the infant's nose or mouth. After his/her head is dried, the infant will receive a cloth cap. Resuscitation will occur in the delivery room and the infant will be wrapped in a blanket and taken to the nursery where he/she will remain in the plastic bag until 1 hour after birth.
  Arms: Resuscitation-torso bag
Procedure: Resuscitation-no plastic bag — Infant will be immediately dried and resuscitated in the delivery room per standard of care. The infant will be wrapped in a blanket and will receive a cloth hat before being taken to the nursery.
  Arms: Resuscitation-no plastic bag

SUMMARY:
The overall hypothesis is that plastic bags used in combination with WHO thermoregulation care will reduce the incidence of hypothermia in preterm/low birth weight and full term infants when compared to routine WHO thermoregulation care alone. Part V is comparing standard WHO thermoregulation practices plus use of a plastic torso wrap to no plastic torso wrap in full term infants from resuscitation to one hour after birth.

DETAILED DESCRIPTION:
Due to delivery rooms without adequate climate controls, even full term infants have high rates of hypothermia in the developing world. This study will compare the rates of hypothermia one hour after birth in full term infants randomized to receive standard WHO thermoregulation care (control group) or standard WHO thermoregulation care without immediate drying plus a plastic bag covering their torsos and lower extremities (intervention group). The axillary temperature of each infant will be taken within 15 minutes of birth at at one hour after birth with removal of the plastic bag. Hyperthermia, room temperature, and death will be recorded throughout the hospitalization for all infants. With an estimated baseline hypothermia rate of 15% and a hypothesized 10% absolute risk reduction (66% relative risk reduction), a sample size of 276 will be used to have a power of 80% and a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age 37 weeks and greater
* Birth weight greater than 2,500gms
* Delivery in the hospital

Exclusion Criteria:

* Infant admitted to the NICU
* Birth weight less than 2,500gms
* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Axillary temperature < 36.5 degrees Celsius | 1-72 hours
  Temperature taken per axilla at one hour after birth. Temperatures 36.0-16.4 will be classified as mild hypothermia, 32.0-35.9 will be classified as moderate hypothermia, and < 32.0 will be classified as severe hypothermia.

SECONDARY OUTCOMES:
Sepsis | Up to 72 hours
  Culture proven or culture negative clinically treated course consistent with sepsis
Death | Up to 72 hours
  Cardiorespiratory failure
Hyperthermia | Up to 72 hours
  Axillary temperature > 38 degrees Celsius per axilla for one minute
Room Temperature | 1-72 hours
  A recording of the room temperature will be obtained with each axillary temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Derived] Belsches TC, Tilly AE, Miller TR, Kambeyanda RH, Leadford A, Manasyan A, Chomba E, Ramani M, Ambalavanan N, Carlo WA. Randomized trial of plastic bags to prevent term neonatal hypothermia in a resource-poor setting. Pediatrics. 2013 Sep;132(3):e656-61. doi: 10.1542/peds.2013-0172. Epub 2013 Aug 26. PMID 23979082